CLINICAL TRIAL: NCT02178930
Title: HealthMap: a Cluster Randomised Trial of Interactive Health Plans and Self-management Support to Prevent Cardiovascular Disease in People With HIV
Brief Title: HealthMap: an Interactive Health Plan Randomised Trial to Prevent Cardiovascular Disease in People With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Klassen (Other)
Collaborators: The Alfred (Other); Monash University (Other); Australasian Society for HIV, Viral Hepatitis and Sexual Health Medicine (Unknown); National Association of People with HIV Australia (Unknown); National Health and Medical Research Council, Australia (Other); Victorian AIDS Council (Unknown); Department of Health & Human Services, State Government of Victoria, Australia (Unknown); Flinders University (Other); Living Positive Victoria (Unknown); NSW Ministry of Health (Unknown); University of Melbourne (Other); Deakin University (Other)
Responsible Party: Sponsor-Investigator, Karen Klassen, Clinical Research Fellow, Monash University
Organization: Monash University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U1111-1150-6489
Record Dates: First submitted 2014-06-29; First posted 2014-07-01 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: HIV; Cardiovascular Disease
Keywords: HIV; cardiovascular disease; self-management; HIV co-morbidities; self-efficacy; coronary heart disease risk; quality of life
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated self management support (Other): The intervention involves the introduction of an interactive chronic disease support platform into doctor-patient consultations, in addition to a self-management support program. Specifically, the intervention comprises the following interlinked components: within consultation engagement; at home exploration; phone and web-based health coaching.
  Interventions: Other: Integrated self management support
- Usual care (No Intervention): The control group will receive usual care from study sites until all study participants have completed 12 months of follow up from their Baseline Visits. At this point access to the study intervention will be expanded to include control sites.

INTERVENTIONS:
Other: Integrated self management support — The intervention comprises a consultation engagement, at home exploration, phone and web-based health coaching.
  Arms: Integrated self management support

SUMMARY:
The purpose of this study is to improve the health status of people living with HIV in Australia. The overall goal is to rigorously evaluate the impact of interactive health plans and self-management support on chronic condition outcomes in people with HIV.

The specific aims are to:

Aim 1: Using a doctor-level cluster randomised trial, evaluate the effect of interactive health plans and self-management support on coronary heart disease risk and other chronic condition outcomes in people living with HIV.

Aim 2: Evaluate patient and health care provider experiences and acceptability of interactive health plans and self-management support.

Aim 3: Evaluate intervention cost-effectiveness and effect on health service utilisation.

DETAILED DESCRIPTION:
Participants will be consenting adults 30 years or older without evidence of cardiovascular disease.The study is a pragmatic cluster randomized controlled trial of a complex health system intervention with doctor as the unit of randomization and individual patient outcomes defined as primary and secondary endpoints. The primary endpoint will be assessed in each participant after 12 months of follow up.The study intervention will consist of a programme specifically designed for the Australian clinical context that helps people with HIV and their health care providers achieve best practice targets for modifiable cardiovascular risk factors. The programme will be available to use during routine consultations to present laboratory results, discuss health priorities and describe goals and actions. Patients will be able to access the interactive health plan from home, with associated additional resources, including online peer support. Phone and online health coaching will be available for prioritised patients wanting to reduce their cardiovascular risk. The primary objective is to determine the effect of the intervention on 10-year risk of non-fatal acute myocardial infarction or coronary heart disease death as estimated by the Framingham risk equation. The secondary objective is to alternative cardiovascular risk scores, individual modifiable cardiovascular risk factors, quality of life, mental health, self- management capacity, process and economic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* •HIV infected adults aged 30 years or over.

  * Receiving ongoing primary HIV and general care at a study site and likely to remain in follow up at that site for 12 months.
  * Willing and able to provide written informed consent.

Exclusion Criteria:

* •Diagnosed cardiovascular disease, consisting of coronary heart disease, stroke or transient ischaemia attack, or peripheral arterial disease.

  * Previous participation in a self-management or coaching program.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
The primary study endpoint is 10-year risk of non-fatal acute myocardial infarction or coronary heart disease death as estimated by the Framingham risk equation | 12 months
  Coronary heart disease Framingham risk equation is obtained from: Wilson P, D'Agostino R, Levy D, Belanger A, Silbershatz H, et al. (1998) Prediction of Coronary Heart Disease Using Risk Factor Categories. Circulation 97: 1837 - 1847.

SECONDARY OUTCOMES:
Cardiovascular risk relative to age as measured by the Joint European Taskforce relative risk tables | 12 months
Cardiovascular risk as estimated by an HIV-specific risk score | 12 months
  (Worm Signe W, Sabin C, Weber R, Reiss P, El Sadr W, et al. (2010) Risk of Myocardial Infarction in Patients with HIV Infection Exposed to Specific Individual Antiretroviral Drugs from the 3 Major Drug Classes: The Data Collection on Adverse Events of Anti-HIV Drugs (D:A:D) Study. The Journal of Infectious Diseases 201: 318-330.)
Smoking status as measured by self-report and verified by urinary cotinine in those describing quitting during the study | 12 months
Fasting total cholesterol and total cholesterol:HDL ratio | 12 months
  (measured by serum assay)
Systolic blood pressure | 12 months
  (using a sphygmomanometer)
Body mass index and waist circumference | 12 months
  Body mass index (calculated by weight in kilograms divided by height in metres squared; these are measured using a scale and stadiometer) and waist circumference (measured using a flexible steel measuring tape)
Proportion of patients achieving Australian cardiovascular risk factor management targets | 12 months
  (http://strokefoundation.com.au/healthprofessionals/ clinical-guidelines/guidelines-for-the-assessment-andmanagement- of-absolute-cvd-risk/)
Quality of life as measured by the AQoL-4D instrument | 12 months
Mental health status as measured by the DASS instrument | 12 months
Self-management capacity as measured by the heiQ instrument | 12 months
Proportion of patients with HIV virological suppression | 12 months
  (Below the lower limit of detection of the assay used )
Proportion of patients achieving HIV quality of care measures | 12 months
Evaluation of the intervention program (intervention arm only) | 12 months
  using a questionnaire designed specifically for this study and using structured interviews.
Health care provider related: Evaluation of the intervention program intervention arm only) | 12 months
  Evaluation of the intervention program (intervention arm only) using a questionnaire designed specifically for this study and using structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Elliott, Principal Investigator — Monash University
Locations (14):
- Australia (14):
  - Fountain Street General Practice, Alexandra, New South Wales
  - Coffs Central Medical Centre, Coffs Harbour, New South Wales
  - CPC Medical Practice, Port Macquarie, New South Wales
  - East Sydney Doctors, Sydney, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Riverside Family Medical Practice, Adelaide, South Australia
  - Alfred Hospital, Melbourne, Victoria
  - Melbourne Sexual Health Centre, Melbourne, Victoria
  - Northside Clinic, Melbourne, Victoria
  - Richmond Hill Medical Centre, Melbourne, Victoria
  - Recreation Medical Centre, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Prahran Market Clinic, Melbourne, Victoria
  - Centre Clinic, Melbourne, Victoria

REFERENCES:
- [Derived] Dodson S, Klassen KM, McDonald K, Millard T, Osborne RH, Battersby MW, Fairley CK, Simpson JA, Lorgelly P, Tonkin A, Roney J, Slavin S, Sterjovski J, Brereton M, Lewin SR, Crooks L, Watson J, Kidd MR, Williams I, Elliott JH. HealthMap: a cluster randomised trial of interactive health plans and self-management support to prevent coronary heart disease in people with HIV. BMC Infect Dis. 2016 Mar 5;16:114. doi: 10.1186/s12879-016-1422-5. PMID 26945746